CLINICAL TRIAL: NCT03415659
Title: A Phase I, Open-label, Single-center, Single/Multiple-dose, Dose-escalation/Dose-expansion Clinical Study on Tolerance and Pharmacokinetics of HWH340 Tablet in Patients With Advanced Solid Tumors
Brief Title: Phase I Clinical Study of HWH340 Tablet in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hubei Biological Medicine Industrial Technology Institute Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HWH340-RFPA 20170821
Record Dates: First submitted 2018-01-16; First posted 2018-01-30 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Advanced Solid Tumors; HRD; BRCA Mutation
Keywords: HWH340; pharmacokinetics; dose-escalation; safety; efficacy; dose-expansion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HWH340 monotherapy (Experimental): HWH340 tablet, oral administration
  Interventions: Drug: HWH340 tablet

INTERVENTIONS:
Drug: HWH340 tablet — 1. single escalating dose study starts from 20 mg as the initial dose until the maximum dose group (520mg) or maximum tolerated dose (MTD) has been reached.
  2. multiple-dose study conducted on oral HWH340 tablet BID. The DLTs evaluating period is 4 weeks and the safety evaluation period lasts till 4 weeks after drug withdrawal.
  3. dose-expansion study conducted on oral HWH340 tablet BID in 2 to 4 dose groups. Patients with BRCA mutation OR HRD will be assigned to 2 cohort in each dose group.

SUMMARY:
This is an open-label, dose-escalation/dose-expansion, phase I clinical trial study to investigate the safety, tolerability, and efficacy of HWH340. In addition, the pharmacokinetic characteristics will also be investigated. Three parts are included in this study.

DETAILED DESCRIPTION:
Part one is a single-dose study on tolerance and pharmacokinetics, in which 21-42 patients with advanced solid tumors would be enrolled. Patients will receive escalating dose groups of HWH340 tablet.

Part two is a multiple-dose study on tolerance and pharmacokinetics. Based on the safety assessment, three or four groups would be chosen to conduct the study. 9-24 patients with advanced solid tumors will be enrolled.

Part three is a dose expansion stage on safety and efficacy. Two to four dose-groups would be chosen to conduct the study. 40-60 patients with advanced solid tumors with BRCA mutation OR homologous recombination deficiency (HRD) will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the advanced solid tumors, which have been histologically and/ or cytologically confirmed.
* Patients with advanced solid tumors refractory to standard therapy or for whom no suitable effective standard therapy exists.
* patients in dose expansion stage must meet the following conditions:
* Group 1: Germline and/or systemic BRCA1/2 mutation;
* Group 2: HRD related gene (except BRCA 1/2) mutation;
* For breast cancer patients, Histologically or cytologically confirmed HER2(-), and received ≤3 prior lines of chemotherapy in advanced or metastatic setting;
* 18 ≤ years of age ≤ 70
* Expected survival time ≥ 6 months
* No serious hematopoietic dysfunction exists. Also, normal function of bone marrow and organs such as heart, lung, liver and kidney are required. Within 14 days prior to inclusion, the patients' laboratory examination results must be within normal limits(under the condition of no extra growth factor or blood transfusion): Blood routine examination: Absolute neutrophil count( ANC) ≥ 1.5 × 109/L),Platelets(PLT) ≥ 100 × 109/L, Hemoglobin(Hb) ≥ 100 g/L;Renal function: Serum creatinine (Cr) ≤1.5×ULN ;Hepatic function: Total Bilirubin ≤1.5×ULN, AST and ALT ≤ 2.5 ×ULN (For patients with liver metastases, AST and ALT ≤ 5 × ULN) ;Electrolytes: normal value ranges (sodium, potassium and calcium);Coagulation function: International Normalized Ratio( INR) ≤1.5, Activated partial thromboplastin time(APTT) ≤ 1.5 × ULN;
* Patients of reproductive potential must agree to practice effective medically approved contraceptive methods during the trial and 6 months afterwards. Women of childbearing potential must have a negative pregnancy test within 7 days prior to screening.
* Subject must fully understand this study, sign informed consent on a voluntary basis , comply with procedures and follow-up examinations as outlined in the protocol and agree to have the gene test.
* Eastern Cooperative Oncology Group (ECOG) performance score ≤ 2 (patients in the multiple-dose study)
* Multiple-dose patients must have no less than one measurable tumor according to RECIST 1.1 criteria.

Exclusion Criteria:

* Subject who has other serious and/or uncontrollable damaged vital organs or unstable systemic disease besides tumors. These diseases include but not limit to uncontrolled diabetes, unstable angina pectoris , cerebrovascular accident or transient cerebral ischemia( within 6 months prior to screening), myocardial infarction (within 6 months prior to screening), congestive heart-failure , uncontrolled high blood pressure, active or uncontrollable infection, hepatic/renal/metabolic disease, serious gastrointestinal disease, any mental disease that may affect study abidance ; or any medical conditions, which in the opinion of the study investigators, places the subject at an unacceptably high risk of toxicities and interfere with the study.
* Subject who has previously been treated with PARP inhibitors, including any related clinical trials, except for HWH340. Subjects in dose expansion stage who have previously received PARP inhibitors (including drug clinical trials), except for patients who have not reached a therapeutic dose with a PARP inhibitor, or patients who have used a PARP inhibitor which is not first-line treatment for ≤ 28 days;
* Subject who has received the treatments of inhibitors of CYP3A3 and/or CYP2D6 within 2 weeks.
* Subject who has received chemotherapy, radiotherapy, endocrinotherapy, biotherapy, immunotherapy, Chinese herbal treatment or other anti-tumor treatment within 4 weeks prior to initiation of this study.In the dose expansion stage, except for patients who have begun bisphosphonate or RANK-L inhibitors with stable dose for bone metastases before enrollment.
* Subject who has participated in other clinical trials or used other investigational drug within 3 weeks prior to initiation of this study.
* Subject who has the autoimmune disease, immunodeficiency disease or surgical history of organ transplantation.
* Positive results of HBsAg, HCV antibody, HIV antibody or Syphilis. Patient who has chronic toxic reaction (≥ CTCAE Grade 2) caused by prophase treatment, except the hair-loss patients.
* Subject who has experienced major surgery and has not been fully rehabilitated within 4 weeks prior to this study.
* Subject who is allergic to the investigational drug or similar drugs, or has the history of allergic disease, or is in allergic constitution.
* History of alcohol addiction or abuse.
* Pregnant /lactating women.
* Subject who has the symptoms of CNS metastases.
* History of gastrointestinal dysfunction and difficulty in swallowing that may influence the drug absorption.
* Subject who has received blood transfusion within 4 weeks prior to the study.
* Subject who attends the study is not on a voluntary basis or cannot comply with the protocol.
* Judged by the investigator, for any reason, that the subject is an unsuitable candidate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2018-03-05 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) and recommended dose (RD) by evaluating the safety and tolerability on single dose | up to 7 days after dosing
  Number of Participants with adverse events
Number of Participants With Laboratory Test Abnormalities on single dose | up to 7 days after dosing
  The laboratory test included: hematology, chemistry, urinalysis, and other tests
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) on multiple dose | up to 30 days after dosing
  Number of Participants with adverse events
Number of Participants With Laboratory Test Abnormalities on multiple dose | up to 30 days after dosing
  The laboratory test included: hematology, chemistry, urinalysis, and other tests

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentrations of platinum (Cmax) | Prior to 0 hour, and 0.5, 1, 2, 4, 8, 12, 36 and 48 hours post dose
  Blood samples are obtained and plasma concentrations of HWH340 are determined using a validated atomic absorption spectrometry method.
Tumor Objective Response Rate（ORR） | on day 42 post dose
  Response and progression is evaluated using internationally accepted response criteria and definitions proposed by the RECIST criteria.
Area under the plasma concentration versus time curve (AUC) | Prior to 0 hour, and 0.5, 1, 2, 4, 8, 12, 36 and 48 hours post dose
  AUC referred to area under the plasma concentration-time curve post dose.
Time for Maximum Observed Plasma Concentration (Tmax) | Prior to 0 hour, and 0.5, 1, 2, 4, 8, 12, 36 and 48 hours post dose
  Blood samples are obtained and plasma concentrations of HWH340 are determined using a validated atomic absorption spectrometry method.
Disease Control Rate (DCR) | through study completion, an average of 1 year
  Response and progression is evaluated using internationally accepted response criteria and definitions proposed by the RECIST criteria.
Objective Response Rate by Investigator | through study completion, an average of 1 year
  Response and progression is evaluated using internationally accepted response criteria and definitions proposed by the RECIST criteria.
Disease control rate | through study completion, an average of 1 year
  Response and progression is evaluated using internationally accepted response criteria and definitions proposed by the RECIST criteria.
Duration of response | through study completion, an average of 1 year
  Response and progression is evaluated using internationally accepted response criteria and definitions proposed by the RECIST criteria.
Best overall response | through study completion, an average of 1 year
  Response and progression is evaluated using internationally accepted response criteria and definitions proposed by the RECIST criteria.
Progression Free Survival | through study completion, an average of 1 year
  Response and progression is evaluated using internationally accepted response criteria and definitions proposed by the RECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: TONG Zhongsheng, Principal Investigator — Professor of Medicine
Locations (1):
- Tianjin medical university cancer insititute & hospital, Tianjin, Tianjin Municipality, China